CLINICAL TRIAL: NCT05886088
Title: National, Multicenter, Randomized, Double-blind, Triple-dummy, Phase III Clinical Trial to Evaluate the Efficacy and Safety of LID104 in the Treatment of Type II Diabetes Mellitus
Brief Title: Efficacy and Safety of LID104 in the Treatment of Type II Diabetes Mellitus
Acronym: DÁLIA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LID104-III-0123
Record Dates: First submitted 2023-05-23; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; Linagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- LID104 (Experimental): The patient must take 1 tablet of LID104 plus 1 tablet of placebo of dapagliflozin and 1 tablet of placebo of linagliptin once a day.
  Interventions: Drug: LID104
- Dapagliflozin (Active Comparator): The patient must take 1 tablet of dapagliflozin plus 1 tablet of placebo of LID104 and 1 tablet of placebo of linagliptin once a day.
  Interventions: Drug: Dapagliflozin
- Linagliptin (Active Comparator): The patient must take 1 tablet of linagliptin plus 1 tablet of placebo of LID104 and 1 tablet of placebo of dapagliflozin once a day.
  Interventions: Drug: Linagliptin

INTERVENTIONS:
Drug: LID104 — Experimental
  Arms: LID104
Drug: Dapagliflozin — Active comparator
  Arms: Dapagliflozin
Drug: Linagliptin — Active comparator
  Arms: Linagliptin

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of LID104 in the treatment of type 2 diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Ability to confirm voluntary participation and agree to all trial purposes by signing and dating the consent form;
* Diagnosis of type II diabetes mellitus, and who did not reach the therapeutic goal of HbA1c with previous dietary, physical exercise and monotherapy with the maximum tolerated dose of metformin at a stable dose in the last 3 months and which, in the Investigator's discretion, may benefit from the addition of the trial drugs.
* Participants with HbA1c ≥ 7.5% and ≤ 10.5% at the screening visit.
* Participants with body mass index ≤ 45 kg/m2

Exclusion Criteria:

* Any clinical observation or laboratory condition finding that is interpreted by the investigating physician as a risk to the participation of the research participant in the clinical trial or presence of uncontrolled chronic disease(s);
* History of alcohol and/or illicit drug use disorder in the last two years;
* Participants who are pregnant, nursing or planning to become pregnant, or female participants of childbearing potential who are not using reliable contraception;
* Participants with known allergy or hypersensitivity to the components of the drugs used during the clinical trial;
* Participants with a current medical history of cancer and/or treatment for cancer in the last five years;
* Participation in a clinical trial protocols in the last 12 months (CNS Resolution 251, of August 7, 1997, item III, subitem J), unless the investigator judges that there may be a direct benefit at the same;
* Type 1 Diabetes Mellitus;
* Fasting glucose above 300 mg/dL;
* Participants who have risk factors for severe volume depletion;
* Participants on dialysis;
* History of metabolic acidosis and/or using medications that may cause lactic acidosis;
* Participants who have had a cardiovascular event (acute myocardial infarction, acute coronary syndrome, recent onset of stable angina, stroke, unstable congestive heart failure requiring change in treatment), who underwent a revascularization procedure or vascular surgery in the six months prior to screening;
* Known heart failure, class III to IV (New York Heart Association);
* Moderate or severe renal insufficiency;
* Participant with altered liver function, defined by serum levels of aspartate aminotransferase, alanine aminotransferase or alkaline phosphatase above three times the upper limit of normal or bilirubin > 1.5 times the upper limit of normal;
* Participants who underwent bariatric surgery in the last two years and/or other gastrointestinal surgeries that may cause chronic malabsorption;
* Medical history of haemoglobinopathies, blood dyscrasia or any other hemolytic disorders;
* Known medical history of pancreatic diseases that may suggest insulin deficiency;
* Known uncontrolled hypothyroidism or hyperthyroidism or thyroid-stimulating hormone (TSH) dosage greater than 1.5 times the reference value;
* Known history of sepsis, hypotension, major surgery, trauma, severe metabolic, endocrine and electrolyte changes or uncontrolled seizures in the six months prior to trial screening, or any other condition that, in the judgment of the investigator, may favor clinically significant alterations in the levels of the enzyme creatine phosphokinase (CPK) or participants with CPK dosages greater than ten times the value considered for normality;
* Participants who started treatment with anti-obesity drugs less than three months ago or with a dose change in the last three months;
* Participants with current and prolonged treatment for more than fifteen days with systemic steroids at the time of informed consent or in the last three months prior to the screening visit;
* Participants on insulin therapy or using oral antidiabetics other than metformin;
* Participants using prohibited medications according to the study protocol.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 597 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | 120 days
  Change from baseline in glycated hemoglobin

SECONDARY OUTCOMES:
Fasting blood glucose | 120 days
  Change from baseline in fasting blood glucose
HbA1c reduction to < 7% | 120 days
  Proportion of participants with HbA1c reduction to < 7%
Treatment failure | Up to 140 days
  Proportion of participants who were discontinued from the study because they needed medication other than the study medication for blood glucose control
Body weight | Up to 140 days
  Change from baseline in body weight
Blood pressure | Up to 140 days
  Change from baseline in blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Investigational site, Hortolândia, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No